CLINICAL TRIAL: NCT06469333
Title: Theories of Working Memory and Consolidation/RECOnsolidation in the Process of Resorption of Certain Post-traumatic Symptoms: Interventional, Randomized Single-center Study
Brief Title: Theories of Working Memory and Consolidation/RECOnsolidation in the Process of Resorption of Post-traumatic Symptoms.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lorraine (Other)
Responsible Party: Principal Investigator, Christine Rotonda, Methodologist/Epidemiologist Head of Research Unit, Pierre Jane Centre, University of Lorraine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-A00296-41
Record Dates: First submitted 2024-06-05; First posted 2024-06-21 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Working Memory; Consolidation/Recconsolidation Memory; Eye Movement Desensitization and Reprocessing; Alterning Bilateral Stimulation; Stress Disorders, Post-Traumatic; Intrusive Memories; Vividness; Emotivity
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Eye Movements

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): The participant is asked to concentrate on the image or, failing that, the sensory representation representing the worst aspect of the targeted intrusive thought for 10 seconds, and to stare at the black computer screen.
- Eye movements (EM) (Experimental): The participant is asked to focus on the image or, failing that, the sensory representation representing the worst aspect of the targeted intrusive thought for 10 seconds and visually follow the horizontal displacement of a white dot (Ø 1cm) on the black screen at a constant speed of 1.2 Hz. This speed, implying the displacement of 1.2 left-right-left cycles per second, targets the saturation of working memory.
  Interventions: Behavioral: Eye movements (EM)
- Eye movements and auditory stimulations (EM+AS) (Experimental): The participant will have to concentrate on the image or, failing that, the sensory representation representing the worst aspect of the targeted intrusive thought for 10 seconds and follow the horizontal displacement of a white dot on the computer screen, while simultaneously perceiving the auditory "beep" tones in the headphones provided. These tones will be at a rate of 1.2 Hz (i.e. 1.2 left ear-right ear-left ear alternations per second).
  Interventions: Behavioral: Eye movements (EM); Behavioral: Auditory stimulations
- Eye movements, auditory stimulations and tactile stimulations (EM+AS+TS) (Experimental): The participant is asked to concentrate on the image or, failing that, the sensory representation representing the worst aspect of the targeted intrusive thought for 10 seconds, and to follow the horizontal displacement of a white dot on the computer screen and simultaneously perceive the "beeps", as well as the tactile self-stimulations applied at a constant speed of 1.2Hz (i.e. 1.2 left-right-left tapping cycles per second).
  Interventions: Behavioral: Eye movements (EM); Behavioral: Auditory stimulations; Behavioral: Tactile stimulations

INTERVENTIONS:
Behavioral: Eye movements (EM) — The participant focuses on the intrusive thought and visually follows the horizontal movement of a white dot (Ø 1 cm) on the black computer screen 8 times for 24 seconds.
  Arms: Eye movements (EM); Eye movements and auditory stimulations (EM+AS); Eye movements, auditory stimulations and tactile stimulations (EM+AS+TS)
Behavioral: Auditory stimulations — The participant focuses on the intrusive thoughts and hears the auditory "beeps" through the headphones provided 8 times for 24 seconds.
  Arms: Eye movements and auditory stimulations (EM+AS); Eye movements, auditory stimulations and tactile stimulations (EM+AS+TS)
Behavioral: Tactile stimulations — The participant focuses on the intrusive thought and applies tactile self-stimulation 8 times for 24 seconds.
  Arms: Eye movements, auditory stimulations and tactile stimulations (EM+AS+TS)

SUMMARY:
EMDR is a psychotherapeutic approach recommended by the World Health Organization (WHO) for the treatment of disorders such as post-traumatic stress disorder, anxiety, depression and, more generally, psychological distress. In all these disorders, intrusions are one of the symptoms leading to intense emotional distress. EMDR therapy, by making intrusions less emotional and less present in the mind (i.e. less vivid), would reduce psychological distress. This symptomatological reduction would be made possible by the therapist's application of alternating bilateral visual (rapid eye movements following a point from left to right), auditory (tones emitted alternately in the right ear and then in the left ear) and/or tactile (tapping with fingers on the left and right shoulders alternately) stimulations administered while the patient concentrates on his or her intrusive thoughts. Accordingly, the aim of this research is to investigate the efficacy of self-administration of Alternating Bilateral Stimulations (ABS), on the emotional intensity (emotionality) associated with negative intrusive thoughts (or intrusions).

DETAILED DESCRIPTION:
Intrusive thoughts (or intrusions) are recognized as being particularly vivid and emotionally "charged", and constitute one of the transdiagnostic symptoms of numerous disorders such as Post Traumatic Stress Disorder (PTSD), anxiety and depression.

Numerous studies have demonstrated that it is now possible to modulate the persistence of intrusions in memory, as well as their emotional impact, through Eye Movement Desensitization and Reprocessing (EMDR) therapy. EMDR is based on the administration of visual, auditory (sound) or sensory (tapping) Alternating Bilateral Stimulations (ABS). These ABS, which can be self-administered by the patient during the Memory Activation (MA) of an intrusive thought, would reduce the emotionality and vividness of the intrusive symptoms and decrease the associated physiological reactivity.

Recent research claims that the mechanisms of action of ABS involve a joint articulation of both neurobiological (Memory Consolidation/Reconsolidation (M-C/R) and psychological (Working Memory (WM)) theories.

Memory consolidation refers to the transfer of a newly acquired memory trace into WM (fragile and susceptible to forgetting) and its stabilization in Long-Term Memory (LTM). Consolidation involves two processes. The first, synaptic consolidation, requires the triggering of molecular processes operating within a time window of between 10 minutes and 6 hours. The second, called systemic consolidation, can extend over years and takes place mainly during the sleep cycle. Reconsolidation implies that an intrusion, when activated in WM, becomes labile again and must subsequently be consolidated again (reconsolidated) in LTM. A permanent memory can thus be revived, then degraded, notably by the administration of ABS likely to interfere with its reconsolidation in memory.

Working memory (WM) refers to a memory system that enables the temporary retention and processing of information needed to perform complex cognitive tasks. capacity is limited. In fact, the competition of two simultaneous tasks (e.g. BAS administration during the memory activation (MA) of an intrusive thought) implies, in a consequential way, an alteration in its storage performance, as well as a decrease in the emotional load associated with the intrusion. In other words, while WM remains the strongest lead to date, it can only be considered in conjunction with M-C/R theory.

From a clinical/experimental protocol point of view, this link implies compliance with a number of criteria. The first is the temporal criterion for ABS administration (between 10 minutes and 6 hours post-MA), as well as the quantitative criterion relating to the number of MAs (not to exceed 4 MAs). In other words, the application of an interventional methodology that does not meet all these criteria (i.e., administration of ABS performed outside the M-C/R time window and repeated MA of the same intrusion) would induce the involvement of a third process, namely the extinction process. In one study, the application of an extinction protocol performed within the consolidation window (a paradigm known as Retrieval Extinction (P-R/E)) also induced a modification of the initial memory trace. It would therefore seem appropriate to consider the adoption of a tri-processual integrative model involving the joint articulation of Working Memory (WM), Memory Consolidation/Reconsolidation (C/R-M) and the Retrieval Extinction Paradigm (P-R/E). This is why we propose to study, in this research , the role of the application of this tri-processual theoretical modeling on the emotionality and vividness associated with intrusions, as well as on their psychophysiological and psychopathological consequences. Through the use of new technologies, these methodologies could complement conventional psychotherapeutic treatments which, through the self-administration of ABS, could add up and, in fact, potentiate the effectiveness of psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Present symptoms of acute stress (score between 22 and 35 on the Impact Event Scale-Revised, IES-R) and/or PTSD (higher score or equal to 36 on the IES-R), but at least present moderate to high psychological distress (score equal to or greater than 8 on the Kessler Abbreviated Psychological Distress Scale, K6);
* Being in need of psychotherapeutic follow-up but not having started it yet;
* Be aged between 18 and 65 years inclusive;
* Speak and write French (be able to understand information and complete questionnaires independently);
* Have good vision (being able to follow the movement of a white point on a screen);
* Have good hearing and tactile abilities (being able to perceive auditory and tactile tones);
* Have a computer equipped with a webcam;
* Be informed and sign informed consent.

Exclusion Criteria:

* Be an adult protected under guardianship or curatorship;
* Be a person subject to a judicial safeguard measure;
* Present a lack of autonomy implying an impossibility in terms of administering questionnaires and filling out questionnaires;
* Have a vision defect implying an impossibility of visual tracking of a white dot;
* Present a hearing defect and/or tactile abilities implying an impossibility of perception;
* Have a neurological condition constituting measurement biases (muscular dysfunctions, perceptual dysfunctions, etc.);
* Suffer from psychotraumatic and dissociative disorders of complex type (respectively evaluated with regard to the anamestistic data of the patients and with a score greater than 25 on the dissociative experiences scale (Dissociative Experiences Scale, DES);
* Do not present psychological distress (score less than 8 on the Kessler Abbreviated Psychological Distress Scale, K6) ;
* Have a drug or alcohol dependence;
* Benefit from ongoing psychotherapeutic monitoring;
* Have already benefited from psychotherapeutic follow-up or have participated in studies in the last 6 months, both involving EMDR therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Measurement of emotionality associated with an intrusive thought | Before and after the experimental phase (7 days after Day 1), The first day after the experimental phase and one night's sleep (comprising 4 to 6 sleep cycles with an average duration of 90 minutes ), through study completion (21 days after D1)
  Emotionality will be assessed using the Subjective Units of Disturbance Scale (SUDS), which ranges from 0 ("no distress at all") to 10 ("maximum distress") and provides a subjective assessment of the disturbance associated with the intrusive thought.

SECONDARY OUTCOMES:
Assessment of the vividness of the intrusion | Before and after the experimental phase (7 days after Day 1), The first day after the experimental phase and one night's sleep (comprising 4 to 6 sleep cycles with an average duration of 90 minutes ), through study completion (21 days after D1)
  Vividness will be assessed via an analogous 11-point numerical scale ranging from 0 ("not vivid at all") to 10 ("extremely vivid"). This measure is frequently used in experimental research involving the application of a double task
Psychological distress | At day 1 (D1), before the experimental phase (7 days after Day 1), The first day after the experimental phase and one night's sleep (comprising 4 to 6 sleep cycles with an average duration of 90 minutes ), through study completion (21 days after D1)
  Psychological distress will be assessed using Kessler's Abbreviated Scale of Psychological Distress. This 6-item scale assesses the frequency of occurrence over the past month of anxiety-depressive emotional states and non-specific psychological distress. On a 5-point scale ranging from 0 "never" to 4 "all the time", the subject is asked to indicate how often he or she felt "nervous", "hopeless", "restless or out of place", "so depressed that nothing could make him or her smile", "that everything was an effort" and that he or she was "good for nothing". The total score obtained ranged from 0 to 24. According to the authors, a total score between 0 and 7 indicates low-intensity distress, a score of 8 to 12 indicates moderate distress, and a score of 13 or above indicates severe psychological distress.
Intrusion symptoms | At day 1 (D1), the first day after the experimental phase and one night's sleep (comprising 4 to 6 sleep cycles with an average duration of 90 minutes ) , through study completion (21 days after D1).
  Symptoms of intrusion will be measured using the Impact of Event Scale-Revised (IES-R). The IES-R is a 22-item scale measuring symptoms of intrusion (dreams about the event), avoidance/blunting (efforts to avoid reminders of the event) and hyperactivation (hypervigilance) in relation to a specific life-threatening event. The subject is asked to indicate on a 5-point Likert scale, from 0 "Not at all" to 4 "Extremely", how upset he or she may have been by difficulties relating to a specific stressful event over the past 7 days. The authors agree that a total score of 22 suggests the presence of acute stress, and a score of 36 indicates the presence of PTSD.
Nature, impact and severity of insomnia | the first day after the experimental phase and one night's sleep (comprising 4 to 6 sleep cycles with an average duration of 90 minutes )
  Insomnia will be measured by the Insomnia Severity Index (ISI) self-report questionnaire. This questionnaire consists of 7 items rated on a 5-point Likert scale. The total score, ranging from 0 to 28, is obtained by adding the scores of the 7 items. A high score of 28 or more indicates severe insomnia; a score of 15 to 21 indicates moderate insomnia; a score of 8 to 14 indicates sub-clinical insomnia. Finally, a score of 7 or less means no insomnia.

OTHER OUTCOMES:
Heart rate variability (HRV) | Before and during the experimental phase (7 days after Day 1)
  Physiological measurement will be carried out by collecting Heart Rate Variability (HRV) using the CardiaSens system (http://www.i-virtual.fr/). RMSSD will be measured using the CardiaSens software integrated into the data collection system, before and after participants complete the questionnaires. Frequency and non-linear analyses of the VFC will also be carried out to complete the understanding of parasympathetic regulation in terms of flexibility and complexity.
Dissociative disorder | At day 1 (D1)
  The presence of a dissociative disorder is assessed using the Dissociative Experiences Scale (DES). This self-administered questionnaire will be used to verify the non-inclusion criterion. Comprising 28 items, this scale measures the frequency of various dissociative symptoms in the respondent's daily life. Two factors are explored: episodes of automatic dissociation linked to the pilot (e.g., associated with different types of cognitive failure) and episodes of defensive dissociation that may act as defensive mechanisms, particularly in traumatized individuals (e.g., avoidance of a memory linked to a traumatic event). The total score is obtained by adding up the scores of the 28 items and dividing by 28, the resulting score ranging from 0 to 100. A high score, greater than or equal to 25, means that patients are more likely to have a dissociative disorder.
Alcohol and drug consumption and the presence of psychotic disorders | At day 1 (D1)
  The Mini International Neuropsychiatric Interview (M.I.N.I.) items assessing alcohol and drug use and the presence of psychotic disorders (pages 16 to 22) will be used to assess the absence of the participants' non-inclusion criteria, namely "drug or alcohol dependence" and "psychiatric history (psychosis type)". The M.I.N.I. has been designed as a brief, structured diagnostic interview for the major psychiatric disorders of the DSM-V.

CONTACTS AND LOCATIONS:
Locations (1):
- Umr U1319 Inspiire, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No